CLINICAL TRIAL: NCT06913244
Title: Long-Term Multidisciplinary Physiotherapy for Breast Cancer Survivors: Evaluation of the 12-Month Effectiveness on Pain, Upper Limb Function, and Cancer-Related Fatigue in a Multi-Center, Parallel-Group Randomized Controlled Trial
Brief Title: Long-Term Multidisciplinary Physiotherapy for Breast Cancer Survivors: A Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al Hayah University In Cairo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BCPhysio2025-01
Record Dates: First submitted 2025-03-30; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Breast Cancer Female
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be randomized (stratified if necessary) to one of two groups-an intervention group receiving the multidisciplinary physiotherapy program and a control group receiving standard care. Both groups will be followed for 12 months to assess clinical and patient-reported outcomes.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the interventions, participants, care providers, and investigators will be aware of the treatment allocation; however, outcome assessors will remain blinded to reduce assessment bias.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multidisciplinary Physiotherapy Program (Experimental): Participants in this arm will undergo a standardized multidisciplinary physiotherapy program consisting of:
  Specific Exercise Therapy: 30-60-minute sessions conducted thrice weekly for 8 weeks (supervised) with subsequent home-based maintenance.
  Manual Therapy: 20-30-minute soft-tissue mobilization sessions twice weekly for 4 weeks.
  Education: Three sessions (in-person and online) focusing on pain neuroscience and self-management strategies.
  Mind-Body Interventions: 40-minute yoga or tai chi sessions once weekly for 6 weeks.
  Interventions: Behavioral: Multidisciplinary Physiotherapy Program (MD Physio)
- Control - Standard Care (Active Comparator): Participants in the control arm will receive "standard care" as currently practiced. This includes routine follow-up and basic physiotherapy advice typically provided to breast cancer survivors without the structured, multidisciplinary program.
  Interventions: Behavioral: Standard Physiotherapy Care

INTERVENTIONS:
Behavioral: Multidisciplinary Physiotherapy Program (MD Physio) — A comprehensive program that integrates:
  Specific Exercise Therapy: Supervised stretching and strengthening sessions (30-60 minutes/session, 3× per week for 8 weeks) followed by a prescribed home-based maintenance regimen.
  Manual Therapy: Targeted soft-tissue mobilization and myofascial release (20-30 minutes/session, twice per week for 4 weeks).
  Education Sessions: Three sessions (both in-person and online) covering pain neuroscience and self-management techniques.
  Mind-Body Interventions: Weekly 40-minute sessions of yoga or tai chi for 6 weeks.
  Arms: Multidisciplinary Physiotherapy Program
Behavioral: Standard Physiotherapy Care — Routine care involves standard follow-up with basic physiotherapy advice as currently provided to breast cancer survivors. This serves as the active comparator in the trial.
  Arms: Control - Standard Care

SUMMARY:
This multi-center randomized controlled trial (RCT) evaluates the long-term (12-month) effectiveness of a standardized multidisciplinary physiotherapy program versus standard care on persistent pain, upper limb (UL) dysfunction, and cancer-related fatigue (CRF) in breast cancer survivors. The study also examines improvements in quality of life and psychological well-being. The standardized intervention combines specific exercise therapy, manual therapy, education, and mind-body interventions and is designed to produce sustained benefits beyond the acute rehabilitation phase.

DETAILED DESCRIPTION:
Breast cancer survivors frequently experience persistent pain, upper limb dysfunction, and CRF well into the survivorship phase, even after completion of acute treatment. Despite various studies evaluating individual interventions, long-term outcomes remain inconclusive due to heterogeneity and short follow-up durations (Devoogdt & De Groef, 2024; McNeely et al., 2010). This study proposes a standardized, multidisciplinary physiotherapy program that integrates:

Specific Exercise Therapy: Structured stretching and strengthening sessions targeting UL mobility and overall fitness (30-60 minutes per session, three times weekly for 8 weeks under supervision, followed by individual home-based maintenance).

Manual Therapy: Targeted soft-tissue mobilization and myofascial release (20-30 minutes per session, twice weekly for 4 weeks).

Education: In-person and online sessions on pain neuroscience and self-management delivered in three sessions.

Mind-Body Interventions: Yoga or tai chi sessions (40 minutes per session, once weekly for 6 weeks).

In this multi-center, parallel-group design, 146 women (aged 18-65) who have undergone breast cancer surgery (with or without axillary lymph node dissection) and completed acute treatment, yet experience persistent sequelae, will be enrolled. Participants will be randomized into two groups: one receiving the multidisciplinary physiotherapy program and the other receiving standard care (routine follow-up with basic physiotherapy advice).

Primary outcomes are measured by changes in pain intensity (VAS), upper limb function (DASH), and CRF (FACIT-Fatigue) at baseline, 3, 6, and 12 months. Secondary outcomes include quality of life (SF-36) and psychological well-being (HADS).

Data will be analyzed using intention-to-treat principles with mixed-effects regression models to adjust for baseline covariates. This study will provide high-quality long-term data to potentially standardize physiotherapy care protocols for breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

Women aged between 18 and 65 years. History of breast cancer surgery (with or without axillary lymph node dissection).

Completed acute cancer treatment (surgery, chemotherapy, and/or radiation) at least 6 months prior to enrollment.

Currently in the survivorship phase, with no active evidence of disease.

Experiencing persistent sequelae related to treatment, such as:

Moderate to severe pain (e.g., VAS score ≥ 30 on a 0-100 scale), and/or Upper limb dysfunction, and/or Cancer-related fatigue (as measured by FACIT-Fatigue). Able to understand and provide written informed consent.

Exclusion Criteria:

Diagnosis of recurrent or metastatic breast cancer. Currently receiving active cancer treatment (chemotherapy, radiation for active disease, or immunotherapy).

Participation in another interventional trial targeting pain or rehabilitation within the past 3 months.

Presence of severe comorbidities (e.g., uncontrolled cardiovascular disease, severe orthopedic or neurological conditions) that would preclude safe participation in physiotherapy.

Any physical or psychological condition that, in the opinion of the investigator, would interfere with participation or adherence to the study protocol (e.g., severe cognitive impairment).

Pregnancy or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2025-04-23 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity (Visual Analog Scale - VAS) | Baseline, 3 months, 6 months, and 12 months post-intervention.
  The VAS is a 0-100 scale used to measure patient-reported pain intensity, where 0 indicates no pain and 100 indicates the worst imaginable pain.
Upper Limb Function (DASH Questionnaire) | Baseline, 3 months, 6 months, and 12 months post-intervention.
  The Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire assesses upper limb function and symptoms with higher scores indicating greater disability.
Cancer-Related Fatigue (FACIT-Fatigue) | Baseline, 3 months, 6 months, and 12 months post-intervention.
  The FACIT-Fatigue scale is a validated tool used to assess the level of fatigue experienced by patients, with lower scores representing greater fatigue.

SECONDARY OUTCOMES:
Quality of Life (SF-36 Health Survey) | Baseline, 3 months, 6 months, and 12 months post-intervention.
  The SF-36 assesses overall health status across multiple domains, providing a composite measure of quality of life.
Psychological Well-Being (Hospital Anxiety and Depression Scale - HADS) | Baseline, 3 months, 6 months, and 12 months post-intervention.
  The HADS is used to evaluate anxiety and depression levels in participants, with higher scores indicating greater psychological distress.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Al Hayah University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No